CLINICAL TRIAL: NCT05828654
Title: Adapting Peer Connect to Train Lay Navigators in Delivering Psychosocial Support to Older Adults With Cancer
Brief Title: Intervention to Address Psychosocial Needs Among Socially Disadvantaged Older Adults With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2240
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hematological Disorder
Keywords: Socially Disadvantaged; older; Psychosocial; need
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Community representatives
  Interventions: Behavioral: Focus Group Discussions and Semi-structured Interviews; Behavioral: Training community lay navigators

INTERVENTIONS:
Behavioral: Focus Group Discussions and Semi-structured Interviews — Community representatives will be asked to participate in either 1:1 semi-structured interviews with a research staff member or to engage in focus group discussions with other community members. These interviews and discussions will gather broad perspectives on resource and training needs for community lay navigators and inform the adaptation of existing Peer Connect training materials
Behavioral: Training community lay navigators — Lay navigators identified from among the recruited community representatives will be trained either in-person or virtually by research staff members in motivational interviewing and other strategies to provide psychosocial support to older socially disadvantaged adults with cancer. For community lay navigators and inform the adaptation of existing Peer Connect training materials.

SUMMARY:
The purpose of this study is to convene a group of diverse North Carolina-based community representatives (patients, caregivers, leaders of faith-based organizations, social workers, and patient navigators) to inform the adaptation of materials used to train lay navigators in the delivery of psychosocial support interventions tailored to older socially disadvantaged adults with cancer.

DETAILED DESCRIPTION:
This behavioral study will explore community representatives' perspectives on the resources and training needed to support the development of a lay navigation program tailored to older socially disadvantaged adults with cancer.

It was hypothesized that diverse community representatives could inform the adaptation of training materials (Peer Connect) and subsequent training of community lay navigators, who will then be positioned to address the psychosocial needs of older adults with cancer

ELIGIBILITY:
Inclusion criteria to participate in the study:

1. Patients aged 65 and older diagnosed with hematological cancer for at least one year with stable disease
2. Community representative 18 years or older who also identifies as at least one of the following:

   1. Cancer caregivers
   2. Social workers, social work students, or patient navigators Community leader (e.g., leader of a faith-based organization)
   3. Previously or currently serve as a lay navigator/peer supporter, community health worker, or coach
   4. Have personal experience with any of the following (being Black race, previously or currently facing socioeconomic challenges, or living in a rural community)
   5. Patient or community representative who is Able to understand and speak in English

Exclusion Criteria

All participants meeting any of the following exclusion criteria at enrollment will be excluded from the study:

1. Inability to read and speak English
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent

Exclusion Criteria

All participants meeting any of the following exclusion criteria at enrollment will be excluded from the study:

1. Inability to read and speak English
2. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Adaptation of the existing Peer Connect training materials- interviews | 12 months
  Through semi-structured interviews, feedback will be qualitatively collected from community representatives to guide the adaptation and further refinement of lay navigator training materials.
Adaptation of the existing Peer Connect training materials- focus group discussions | 12 months
  Through focus group discussions, feedback will be qualitatively collected from community representatives to guide the adaptation and further refinement of lay navigator training materials.

SECONDARY OUTCOMES:
Training community lay navigators- training sessions | 12 months
  The ability to train community lay navigators using the newly adapted training content- training sessions will be assessed by the number of training sessions completed by lay navigators and the research staff, allowing for sharing of broad perspectives on training methods, content, and delivery.
Training community lay navigators - semi-structured interviews | 12 months
  The ability to train community lay navigators using the newly adapted training content will be assessed through qualitative semi-structured interviews with lay navigators and the research staff, allowing for sharing of broad perspectives on training methods, content, and delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Shakira Grant, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials